CLINICAL TRIAL: NCT03543787
Title: Strengthening Referral Networks for Management of Hypertension Across the Health System (STRENGTHS)
Acronym: STRENGTHS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Moi University (Other)
Collaborators: Indiana University (Other); Duke University (Other); Icahn School of Medicine at Mount Sinai (Other); Purdue University (Other); University of Texas at Austin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1U01HL138636-01 (NIH)
Record Dates: First submitted 2017-12-19; First posted 2018-06-01 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Hypertension
Keywords: Referral networks; low and middle income countries; PRECEDE-PROCEED; implementation research; hypertension; cardiovascular disease; process evaluation
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: PRECEDE-PROCEED implementation research framework; 2-arm cluster randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Health IT and Peer Support Intervention (Active Comparator): Utilise electronic decision support, tracking of referral list and Peer facilitation for referral completion
  Interventions: Combination Product: Health IT and Peer Support Intervention
- Non intervention group (No Intervention): 2014 - 2018 MoH referral protocol

INTERVENTIONS:
Combination Product: Health IT and Peer Support Intervention — Health IT will support referral system by establishing 1) communication between healthcare providers and peer navigators 2) decision support for clinician to facilitate appropriate referrals 3) tracking of referred patients real-time 4) dashboards to monitor key evaluation metrics.
  Peer Support intervention: peer navigators at each level of the referral network will ensure 1) referral adherence by link clinicians and patients 2) health system navigation 3) psychosocial support: leverage their shared disease experience to help patients overcome barriers to health seeking behaviour.
  Arms: Health IT and Peer Support Intervention

SUMMARY:
"STRENGTHS" is a transdisciplinary implementation research study, guided by the PRECEDE-PROCEED framework, to address the challenge of improving hypertension control in low-resource settings. The investigators propose to test the hypothesis that referral networks strengthened by an integrated health information technology and peer support intervention will be effective and cost-effective in improving hypertension control among patients in western Kenya. The investigators hypothesise that the integrated Health information Technology and Peer Support intervention will facilitate seamless referral of hypertensive patients across the different levels of the health system compared to usual care, leading to improvement in blood pressure. If proven to be successful, STRENGTHS can serve as a model for improving referral of patients upstream and downstream in health systems worldwide.

DETAILED DESCRIPTION:
Hypertension is a major risk factor for cardiovascular disease, and 80% of global mortality due to cardiovascular diseases occurs in low- and middle-income countries. In low income countries, lack of coordination between different levels of the health system threatens the ability to provide the care necessary to control hypertension and prevent cardiovascular disease related morbidity. Strong referral networks have improved health outcomes for chronic disease in a variety of settings. Health information technology and peer-based support are two strategies that have improved care coordination and clinical outcomes. However, their effectiveness in strengthening referral networks to improve blood pressure control and reduce cardiovascular disease risk in low-resource settings is unknown.

The Academic Model Providing Access to Healthcare (AMPATH) partners with the Kenya Ministry of Health to provide care for non-communicable chronic diseases (NCDs), including hypertension at all levels of the health system. The Kenya Ministry of Health Sector Referral Strategy 2014-2018 calls for improving the referral system at every level of the health system. AMPATH has piloted both health information technology and peer support for NCDs, and both strategies are feasible in this setting. However, the impact of integrating Health information technology and peer support to strengthen referral networks for hypertension control is unknown.

The proposal's objective is to utilise the PRECEDE-PROCEED framework to conduct trans-disciplinary, translational implementation research focused on strengthening referral networks for hypertension control. The central hypothesis is "Health Information Technology integrated with peer support will be effective and cost-effective in strengthening referral networks, improving blood pressure control, and reducing cardiovascular risk among hypertensive patients in western Kenya." The investigators hypothesise that Health information technology(HIT) and peer support(PS) will synergistically address barriers to hypertension control at the patient, provider and health system levels. The investigators further hypothesise that changes in referral network characteristics may mediate the impact of the intervention on the primary outcome, and that baseline referral net-work characteristics may moderate the impact of the intervention. To test these hypotheses and achieve the overall objective, STRENGTHS has the following specific aims:

Aim 1: Conduct a baseline needs and contextual assessment for implementing and integrating HIT and PS to strengthen referral networks for hypertension control, using a mixed-methods approach, including: observational process mapping and gap assessment; baseline referral network analysis; and qualitative methods to identify facilitators, barriers, contextual factors, and readiness for change.

Sub-Aim 1.1: Use data from the aim 1 to develop a contextually and culturally appropriate intervention to strengthen referral networks for hypertension control using a participatory, iterative design process. Conduct pilot acceptability and feasibility testing of the intervention.

Aim 2: Evaluate the effectiveness of HIT and PS for hypertension control by conducting a two-arm cluster randomized trial comparing: 1) usual care vs. 2) referral networks strengthened with an integrated HIT-PS intervention. The primary outcome will be one-year change in systolic blood pressure and a key secondary outcome will be cardiovascular risk reduction.

Sub-Aim 2.1: Conduct mediation analysis to evaluate the influence of changes in referral network characteristics on intervention outcomes, and a moderation analysis to evaluate the influence of baseline referral net-work characteristics on the effectiveness of the intervention.

Sub-Aim 2.2: Conduct a process evaluation using the Saunders framework, evaluating key implementation measures related to fidelity, dose delivered, dose received, recruitment, reach, and context.

Aim 3: Evaluate the incremental cost-effectiveness of the intervention, in terms of costs per unit decrease in SBP, per percent change in CVD risk score, and per disability-adjusted life year (DALY) saved.

This research project will add to the existing knowledge base on innovative and scalable strategies for strengthening referral networks to improve control of NCDs in lower-MICs. If proven to be effective, it has the potential to be a scalable model for other low-resource settings globally.

ELIGIBILITY:
Inclusion Criteria:

* >= 18 yrs
* Enrolled in AMPATH CDM Program
* meet criteria for referral up or down the network

  * Patients with complicated hypertension meet criteria for referral up the network, defined as patients with hypertension who remain uncontrolled (SBP >= 140 or DBP >= 90) on 3 or more anti-hypertensive medications, who have signs or symptoms of end-organ damage, or who have suspected secondary causes of hypertension (age <35 years, HIV, or pregnancy)
  * Patients with stable, uncomplicated hypertension meet criteria for referral down the network, defined as controlled BP (SBP < 140 and DBP < 90) for 3 or more consecutive visits and no evidence of new end-organ damage

Exclusion Criteria:

* acute illness requiring immediate medical attention
* terminal illness
* inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1600 (Actual)
Dates: Start 2020-01-17 (Actual); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in one year systolic blood pressure as measured in clinic | 1 year
  The systolic blood pressure at baseline will be compared to systolic blood after 1 year of follow up. Blood pressure measurements will be averaged from three successive readings taken every 5 minutes in clinic

SECONDARY OUTCOMES:
Change in one year overall Cardiovascular disease (CVD) QRISK2 score | 1 year
  QRISK2 score is a computerised algorithm for predicting the ten-year risk of developing CVD events. The factors that enter into the calculation of the QRISK2 score include: Age 25-84 years, sex, ethnicity, smoking status, diabetes status, family history of coronary artery disease in first degree relatives below the age of 65 years, chronic kidney disease stages 4 and 5, atrial fibrillation, rheumatoid arthritis, cholesterol / high density lipoprotein ratio, systolic blood pressure, body mass index. A score of 10% or more suggest a 10% risk of primary CVD events in ten years and warrants intervention to reduce the risk. It's not used among patients who already have a heart attack or a stroke.
Mortality | 1 year follow up
  Death at the end of the study
Hospitalisation | 1 year of follow up
  Number of self-reported hospital admissions for hypertensive crises or heart failure among participants over one year follow up.
Cardiovascular disease complications | 1 year follow up
  Any cardiovascular complications including Heart failure, Stroke and Acute myocardial infarction
Change in number of CVD risk factors and behaviors as assessed using a standardised screening questionnaire | 1 year
  Baseline risk factor profile compared to profile at 1 year of the various CVD risk factors as assessed using a standardised CVD risk factors and behaviours screening questionnaire
Self reported adherence to hypertension medication as assessed using the Morisky Medication adherence questionnaire | 1 year
  To assess changes in adherence to hypertension medications at one year from baseline as determined using the Morisky medication adherence questionnaire

OTHER OUTCOMES:
Referral network characteristics | 1 year
  To assess the referral densities within the healthcare system.
Referral proces characteristics | 1 year
  To assess referral completion rates within the healthcare system

CONTACTS AND LOCATIONS:
Overall Officials: Constantine O Akwanalo, Principal Investigator — Moi University
Locations (1):
- Constantine Akwanalo, Eldoret, Kenya

IPD SHARING:
Plan to Share IPD: Undecided
After data cleaning and primary analyses, the de-identified data will be available to the scientific community upon formal request made to the AMPATH Research Manager. The data collection instruments will also be available upon request to the AMPATH Research Manager.

REFERENCES:
- [Derived] Naanyu V, Njuguna B, Koros H, Andesia J, Kamano J, Mercer T, Bloomfield G, Pastakia S, Vedanthan R, Akwanalo C. Community engagement to inform development of strategies to improve referral for hypertension: perspectives of patients, providers and local community members in western Kenya. BMC Health Serv Res. 2023 Aug 11;23(1):854. doi: 10.1186/s12913-023-09847-0. PMID 37568172
- [Derived] Thakkar A, Valente T, Andesia J, Njuguna B, Miheso J, Mercer T, Mugo R, Mwangi A, Mwangi E, Pastakia SD, Pathak S, Pillsbury MKM, Kamano J, Naanyu V, Williams M, Vedanthan R, Akwanalo C, Bloomfield GS. Network characteristics of a referral system for patients with hypertension in Western Kenya: results from the Strengthening Referral Networks for Management of Hypertension Across the Health System (STRENGTHS) study. BMC Health Serv Res. 2022 Mar 7;22(1):315. doi: 10.1186/s12913-022-07699-8. PMID 35255913
- [Derived] Mercer T, Njuguna B, Bloomfield GS, Dick J, Finkelstein E, Kamano J, Mwangi A, Naanyu V, Pastakia SD, Valente TW, Vedanthan R, Akwanalo C. Strengthening Referral Networks for Management of Hypertension Across the Health System (STRENGTHS) in western Kenya: a study protocol of a cluster randomized trial. Trials. 2019 Sep 9;20(1):554. doi: 10.1186/s13063-019-3661-4. PMID 31500661

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-09-10): https://cdn.clinicaltrials.gov/large-docs/87/NCT03543787/Prot_SAP_ICF_000.pdf